CLINICAL TRIAL: NCT01678183
Title: Financial Incentives for Medication Adherence
Acronym: FIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Pfizer (Industry); National Bureau of Economic Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BU IRB H-30045; WS2069417 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Monthly Incentive (Experimental): Subjects in this arm will receive a cash incentive each month when they pick up their medications for diabetes, hypertension, and hypercholesterolemia at the pharmacy on time. The intervention is the cash incentive.
  Interventions: Behavioral: Monthly Financial Incentive
- Monthly and Final Incentive (Experimental): Subjects in this arm will receive a cash incentive each month when they pick up their medications for diabetes, hypertension and hypercholesterolemia at the pharmacy on time, as well as an additional financial incentive for each full percentage point of decrease in their hemoglobin A1c over the eight-month course of the study. The two cash incentives are the intervention.
  Interventions: Behavioral: Monthly Financial Incentive; Behavioral: Final Financial Incentive
- Control (No Intervention): These subjects will complete the enrollment process for the study but will be randomized to a group that receives usual care.

INTERVENTIONS:
Behavioral: Monthly Financial Incentive — A cash payment.
  Arms: Monthly Incentive; Monthly and Final Incentive
Behavioral: Final Financial Incentive — One-time payment in cash for each full percentage of hemoglobin A1c decrease over the eight-month period of the study.
  Arms: Monthly and Final Incentive

SUMMARY:
This study is a pilot study. The investigators have designed a randomized, controlled trial of financial incentives in medication adherence, focusing primarily on poorly-controlled diabetes, and secondarily on hypertension, and high cholesterol. Prior work has shown that many patients do not take their medications as prescribed by their doctors. This contributes to increased rates of bad outcomes such as blindness, kidney failure, heart attack, and death. The investigators hypothesize that use of a financial incentive will motivate patients to improve their medication adherence and ultimately their control of their chronic diseases.

The investigators plan to identify patients who get Primary Care at Boston Medical Center who still have high blood sugars more than a year after their diabetes diagnosis, and randomize them to a control arm, or one of two intervention arms. Subjects will be approached at the time of a regularly-scheduled appointment with their Primary Care doctor and offered the opportunity to participate in the study. All subjects who agree to participate in the study will meet with a Clinical Pharmacologist to review their medications in detail, and then undergo randomization. Subjects in the first intervention group will receive a cash incentive for picking up medications for the targeted conditions from the pharmacy each month. Subjects in the second intervention group will receive a cash incentive for picking up medications for the targeted conditions from the pharmacy each month, and a one-time payment at the conclusion of the study based on the amount of hemoglobin A1c decrease. The investigators will enroll a total of 100 subjects in the study, and anticipate an observational cohort of approximately 1,000 patients.

All patients who are eligible for the study but who are not enrolled in the study and have not declined to participate in the study will become the observational cohort for the study. The observational cohort will be used to determine whether randomization to the control arm of the study has a negative, rather than neutral, effect on patients.

At the end of eight months, all subjects will meet with a Visiting Nurse in their home, to have their blood pressure checked and to have their blood drawn so that their blood sugar and cholesterol can be measured. Outcomes to be evaluated include hemoglobin A1c, lipid panel, systolic blood pressure, diastolic blood pressure, self-reported health, microvascular and macrovascular complications, and death.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Speaks English, Spanish, or Haitian Creole
* Established patient in Boston Medical Center Section of General Internal Medicine Primary Care Practice
* Uses Boston Medical Center Pharmacy
* Diagnosed with diabetes for more than one year
* Prescribed medications for diabetes
* Last hemoglobin A1c > 7.9

Exclusion Criteria:

* Pregnant
* History of Brittle Diabetes
* Meets April, 2012 American Diabetes Association criteria for an increased goal hemoglobin A1c

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Improvement in hemoglobin A1c | 8 months
  The investigators will evaluate levels of blood sugar over time as measured by the hemoglobin A1c at the start and end of the study.

SECONDARY OUTCOMES:
Improvement in blood pressure. | Eight months
  The investigators will assess blood pressure measurements at the start and end of the study.

OTHER OUTCOMES:
Lipid levels | Eight months
  The investigators will assess lipid levels at the start and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rourke, MD, Principal Investigator — Boston Medical Center; Amitabh Chandra, Ph.D., Principal Investigator — Harvard Kennedy School, National Bureau of Economic Research; Katherine Baicker, Ph.D., Principal Investigator — Harvard School of Public Health, National Bureau of Economic Research
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States